CLINICAL TRIAL: NCT01961024
Title: Postprandial VLDL-TG Metabolism
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Esben Søndergaard, Post Doc, MD, PhD, University of Aarhus
Other Study IDs: ES-0006
Record Dates: First submitted 2013-09-27; First posted 2013-10-11 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
Keywords: VLDL-TG kinetics; Postprandial state; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — specimen of muscle specimen of adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Type 2 diabetic men
- Age- and weight-matched controls

SUMMARY:
In thise study, we aim to determine the effect of meal fat on VLDL-TG kinetics in type 2 diabetic and healthy subjects matched for BMI in order to elucidate the potential pathophysiological differences in VLDL-TG FA channeling towards oxidation and storage in abdominal and leg subcutaneous adipose tissue. Specifically, we want to measure, by way of fat and muscle biopsies, the quantitative postprandial storage of VLDL-TG FA's in skeletal muscle and adipose tissue in relation to a series of tissue specific proteins and enzymes that might be involved in regulating skeletal muscle and adipose tissue FA storage.

ELIGIBILITY:
Inclusion Criteria:

* Written consent

Exclusion Criteria:

* Known diseases
* Alcohol abuse
* Smoker
* Regular use of medicine

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males with diabetes from the department´s out-patient clinic. Control group of healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
VLDL-TG storage in adipose tissue | 3 hours

SECONDARY OUTCOMES:
18F-THA fractional storage | 6 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology MEA, Aarhus Hospital, Aarhus C, Please Select, Denmark

REFERENCES:
- [Derived] Sondergaard E, Johansen RF, Jensen MD, Nielsen S. Postprandial VLDL-TG metabolism in type 2 diabetes. Metabolism. 2017 Oct;75:25-35. doi: 10.1016/j.metabol.2017.07.002. Epub 2017 Jul 19. PMID 28964326